CLINICAL TRIAL: NCT02310412
Title: A Controlled, In Vivo, Pilot Study to Assess the Recovery and Survival of Radiolabeled Autologous INTERCEPT Treated 7-Day Stored Apheresis Platelet Components in 35% Plasma and 65% InterSol and 7-Day Stored Apheresis Platelet Components in 100% Plasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLI 00099
Record Dates: First submitted 2014-11-10; First posted 2014-12-08 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: INTERCEPT; platelet; pathogen inactivation; platelet components stored; therapeutic efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amicus platelet components (Experimental): The two stages of this pilot study consist of the following: single or double dose platelet apheresis collection, pathogen inactivation with INTERCEPT treatment, storage for 7 days, collection of fresh platelets, radiolabeling, infusion of fresh and stored INTERCEPT treated radiolabeled autologous platelets, and collection of blood samples for assessment of platelet recovery and survival (lifespan). In Stage 1, apheresis platelets will be collected using the Amicus separator and stored for 7 days in 35% Plasma and 65% InterSol
  Interventions: Biological: INTERCEPT treated platelets
- Trima platelet components (Experimental): The two stages of this pilot study consist of the following: single or double dose platelet apheresis collection, pathogen inactivation with INTERCEPT treatment, storage for 7 days, collection of fresh platelets, radiolabeling, infusion of fresh and stored INTERCEPT treated radiolabeled autologous platelets, and collection of blood samples for assessment of platelet recovery and survival (lifespan). In Stage 2, apheresis platelets will be collected using the Trima separator and stored for 7 days in 100% plasma.
  Interventions: Biological: INTERCEPT treated platelets

INTERVENTIONS:
Biological: INTERCEPT treated platelets

SUMMARY:
The objective of this study is to test the hypothesis that INTERCEPT platelet components stored for 7 days retain sufficient viability for therapeutic efficacy. The post-infusion recovery and lifespan of 7-day old INTERCEPT platelet components stored in 35% plasma and 65% InterSol or stored in 100% plasma, will be measured in comparison to "fresh" radiolabeled platelets according to FDA guidance for platelet testing (FDA 1999).

DETAILED DESCRIPTION:
The two stages of this pilot study consist of the following: single or double-dose platelet apheresis collection, pathogen inactivation with INTERCEPT treatment, storage for 7 days, collection of fresh platelets, radiolabeling, infusion of fresh and stored INTERCEPT treated radiolabeled autologous platelets, and collection of blood samples for assessment of platelet recovery and survival (lifespan).

In Stage A, apheresis platelets will be collected using the Amicus separator and stored for 7 days in 35% Plasma and 65% InterSol.

In Stage B, apheresis platelets will be collected using the Trima separator and stored for 7 days in 100% plasma.

Procedures for both stages will be as follows: On Day 0, each healthy volunteer subject has apheresis platelets collected. INTERCEPT treatment will begin on either the day of donation (Day 0) or before the end of the day following donation (Day 1). Platelets will then be stored for 7 days after collection (Day 7). Aliquots for in vitro platelet function will be taken on Day 0/1 after INTERCEPT treatment and Day 7. An aliquot for bacterial detection will be taken on Day 5.

On Day 7, healthy volunteers will return to the laboratory, and 43 mL of blood will be drawn into a syringe containing 9 mL of Anticoagulant Citrate Dextrose Solution, Formula A (ACD-A). Fresh platelets will be prepared from this sample. An aliquot (10-20 mL) of the stored (INTERCEPT treated) platelets will be aseptically removed from each subject's test container. Previously stored (Test) and fresh (Control) platelets will be radiolabeled according to randomization assignment with either 51Cr (≤20 μCi) as sodium radiochromate (Na251CrO4), or 111In (≤15 μCi) as indium oxine, following the labeling and washing procedures outlined by the Biomedical Excellence for Safer Transfusion (BEST) Collaborative. The isotope labels will be determined by a random number table such that equal numbers of fresh and stored (INTERCEPT treated) platelets will be labeled with each isotope. Aliquots of the fresh and stored platelets will be radiolabeled in tubes with the standard techniques. After radiolabeling, the autologous fresh and stored platelets will be simultaneously infused into the subject (approximately 10-30 mL). Negative bacteria detection test and negative pregnancy test for females of childbearing potential are required before infusion.

Blood samples for radioactivity measurements will be drawn at 0 (pre-infusion), 0.5, 1, and 2 hours post-infusion, and then 6 more samples will be drawn 1, 2, 3, 4 (or 6), 7±1, and 10±1 days post-infusion. In addition, when logistically feasible, an additional sample will be obtained 5 days post-infusion (optional).

Radioactivity measurements Samples will be obtained from the radiolabeled fresh and stored platelets before infusion and used as a radioactive standard. By measuring the volume infused, the total dose of radioactivity infused will be calculated. In vitro elution of the label from the transfused platelets will be determined by two elution assessment methods, as well as the in vivo elution of radioactivity from the serial blood samples obtained post-infusion of the labeled platelets.

The standard as well as the subject's whole-blood samples will be corrected for elution and also for the residual activity in the cellular fraction on Day 8. The first four data points post-infusion will be used to calculate in vivo recoveries and survivals after all radioactive corrections have been made. The radioactivity of the samples will be determined by use of a gamma counter. A multiple-hit model, with a computerized program "COST," will be used to estimate the recovery and survival of the radioactively labeled platelets.

ELIGIBILITY:
Inclusion Criteria:

* Age-minimum of 18 years, of either gender
* Normal health status (as determined by the Investigator review of medical history and blood donor physical exam)
* Meet FDA and AABB guidelines for autologous apheresis platelet donation
* Complete blood count (CBC) and serum chemistry values within normal limits
* Pre-donation platelet count of more than 150×109 platelets/L
* Negative blood donor screening test panel for HIV, HBV, HCV, HTLV, syphilis, and WNV
* Male and female subjects of childbearing potential must agree to use a medically acceptable method of contraception throughout the study. A barrier method of contraception must be included, regardless of other methods.
* Signed and dated informed consent form

Exclusion Criteria:

* Clinically significant acute or chronic disease (as determined by the Investigator)
* Pregnant or nursing females
* Male or female subjects of childbearing potential not using effective contraception
* Disease states or conditions that preclude blood donation or apheresis platelet donation per AABB reference standards
* Treatment with aspirin or aspirin containing medications within 7 days of apheresis or treatment with non-steroidal anti-inflammatory drugs (NSAID), anti-platelet agents or other drugs affecting platelet viability within 3 days of apheresis (e.g. ibuprofen or other NSAIDs)
* Smokers using >10 cigarettes/day for the last 3 months
* Splenectomized subjects
* Prior exposure to amotosalen
* History of known hypersensitivity to indium or chromium
* Participation in another clinical study currently or within the past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Post infusion recovery ratio of Test platelets at Day 7 compared to fresh platelets | Day 7
Post infusion lifespan ratio of Test platelets at Day 7 compared to fresh platelets | Day 7
In vitro pH at Day 7 | Day 7
Adverse events, vital signs, hematological profile and serum chemistry profile | Days 0 to 17

SECONDARY OUTCOMES:
Product parameters | Day 7
  Platelet count, platelet dose, mean platelet volume (MPV), morphology score, and volume
Biochemical assessments | Day 7
  glucose, lactate pO2, pCO2, bicarbonate, and lactate dehydrogenase (LDH)
Functional assessments | Day 7
  hypotonic shock response (HSR), extent of shape change (ESC), CD62 (p-selectin)expression, and ATP, % of lysis
Bacterial contamination | Day 7
  A bacterial detection test of the Test component will be performed using the Pall Medical enhanced bacterial detection system (eBDS)